CLINICAL TRIAL: NCT03098108
Title: Concurrent Chemo-proton Radiotherapy With or Without Resection and Spacer Insertion for Loco-regional Recurrence of Previous Irradiated Rectal Cancer: Prospective Phase II Trial
Brief Title: Concurrent Chemo-proton Radiotherapy With or Without Resection and Spacer Insertion for Loco-regional Recurrence of Previous Irradiated Rectal Cancer
Acronym: RECCPT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Hee Cheol Kim, Professor, Samsung Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2016-08-121
Record Dates: First submitted 2017-02-20; First posted 2017-03-31 (Actual); Last update posted 2018-06-28 (Actual); Status verified 2018-06

CONDITIONS: Previously Irradiated Recurrent Rectal Cancer

STUDY DESIGN:
Intervention Model Description: CCPT arm
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CCPT (Experimental)
  Interventions: Radiation: Concurrent chemo-proton therapy

INTERVENTIONS:
Radiation: Concurrent chemo-proton therapy — Proton therapy with simultaneous integrated boost technique Gross tumor volume 70.4 gray (Gy)/ 16 fractions and clinical target volume 44.8 Gy/16 fractions Capecitabine twice a day 825 mg/body square meter
  Other Names: CCPT

SUMMARY:
The investigators conduct this study to evaluate the efficacy and adverse effect of salvage concurrent chemo-proton therapy (CCPT) with or without surgical resection in previously irradiated recurrent rectal cancer.

DETAILED DESCRIPTION:
The obtaining of local control in previously irradiated recurrent rectal cancer is crucial for survival prolongation as well as quality of life of patients. But, it is not easy to get with surgery and/or conventional radiotherapy (RT) because of the limitation of RT dose. Proton therapy has unique advantage showing superior dose distribution focusing tumor escaping surrounding normal tissues using "Bragg-peak".

ELIGIBILITY:
Inclusion Criteria:

* previously diagnosed as rectal cancer and received curative intent treatment
* diagnosed as recurrent rectal cancer either pathology or radiologic exam
* discussed at tumor board and recommend proton therapy
* previous history of pelvic area radiotherapy
* Eastern Cooperative Oncology Group performance status of 0 to 2
* informed consent to present study
* consent to contraception for 6 months during and after study participation
* maintained bone marrow function ( absolute neutrophil count ≥ 1,2 * 109/L, platelet count ≥ 100 * 109/L)
* maintained renal, hepatic function creatinine clearance ≥ 50 mL/minute total bilirubin ≥ 2.2 mg/dl alkaline phosphatase ≥ 192 U/L

Exclusion Criteria:

* Pregnant and/or breastfeeding woman
* Less than 12 weeks of expected survival
* Uncontrolled active co-morbidity

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2017-02-09 (Actual); Primary Completion 2019-10-31 (Estimated); Study Completion 2021-10-31 (Estimated)

PRIMARY OUTCOMES:
local control rate at 3-year | 3-year after CCPT
  Local progression will be defined according to the revised Response Evaluation Criteria in Solid Tumor (RECIST version 1.1)

SECONDARY OUTCOMES:
adverse events | 3 months after CCPT
  Adverse events will be evaluated with the Common Terminology Criteria for Adverse Events (CTCAE) version 4.0.
objective response rate | 1 and 3 months after CCPT
  Local progression will be defined according to the revised Response Evaluation Criteria in Solid Tumor (RECIST version 1.1)
time to local tumor progression | 3-year after CCPT
  Local progression will be defined according to the revised Response Evaluation Criteria in Solid Tumor (RECIST version 1.1)
progression free survival | 3-year after CCPT
  Local progression will be defined according to the revised Response Evaluation Criteria in Solid Tumor (RECIST version 1.1)
Core Quality of life (QOL-C) assessment | Baseline, at last week of CCPT, 1 and 3 months after CCPT
  QOL will be evaluated with European Organisation for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire-Core (QLQ-C) 30.
Colonrectum Quality of life (QOL-CR) assessment | Baseline, at last week of CCPT, 1 and 3 months after CCPT
  QOL will be evaluated with EORTC QLQ- (colonrectum) CR 29.

CONTACTS AND LOCATIONS:
Locations (1):
- Samsung Medical Center, Seoul, South Korea